CLINICAL TRIAL: NCT03223597
Title: Registry of Treatment Outcomes in a Non-study Population of Symptomatic Metastasized Castration Resistant Prostate Cancer (mCRPC) Patients Treated With Radium-223
Brief Title: Registry of Treatment Outcomes of Symptomatic Metastasized Castration Resistant Prostate Cancer Treated With Radium-223
Acronym: ROTOR
Status: Completed | Type: Observational
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: m14ROT
Record Dates: First submitted 2017-04-04; First posted 2017-07-21 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2017-07

CONDITIONS: Prostate Cancer Metastatic; Bone Metastases
Keywords: Radium-223; quality of life; Pain
MeSH Terms: conditions — Pain | interventions — radium Ra 223 dichloride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Radium-223 dichloride — Registry of patients who receive Radium-223.
  Other Names: Xofigo

SUMMARY:
Radium-223 is the 5th treatment for metastasized castration resistant prostate cancer with a proven overall survival benefit. The improved survival of Radium-223 over placebo was demonstrated in the ALSYMPCA trial, which included a miscellaneous patient population both docetaxel pretreated and non-pretreated. This registry aims to describe non-study patients treated with Radium-223 and prospectively evaluate treatment outcomes of patients with and without docetaxel pretreatment. Analgesic use and patient reported pain scores, efficacy of the subsequent therapy and overall survival will be evaluated. Moreover, clinical and explorative serum and blood biomarkers of Radium-223 efficacy will be explored.

DETAILED DESCRIPTION:
Every year approximately 12,000 men are diagnosed with prostate cancer in the Netherlands and approximately 2,400 die of this disease. When prostate cancer is limited to the prostate, patients can be operated or radiated with a curative intention, however, metastasized disease is incurable. Initially, prostate cancer responds to testosterone at castration level and treatment with androgen receptor signaling inhibitors. However, after an average of 24 months, prostate cancer will reach a castration resistant stage (mCRPC), which is associated with high morbidity and mortality. Since the introduction of Docetaxel in 2004, multiple treatments for mCRPC have become available. All these treatments have a proven beneficial effect on quality of life and all expand life expectancy. An important clinical problem is that approximately 50% of older patients are not able or not willing to receive docetaxel treatment. These patients are also not eligible for treatments of docetaxel refractory disease. Therefore, there is a need for effective treatments with little site effects.

In the phase 3, ALSYMPCA study 921 patients were randomized between Rad-223 (Xofigo®) and placebo in a 2:1 distribution1. Patients with symptomatic bone metastases, limited lymph node involvement, adequate bone marrow, kidney and liver functions were included in this trial. Patients were previously treated with docetaxel or could not receive docetaxel, declined docetaxel or docetaxel was not available. At a planned interim analysis after 538 deaths, the primary end point overall survival (OS) was 14.9 months in the Radium-223 treated arm and 11.3 months in the placebo arm (HR 0.70; 95% CI 0.58-0.83). All secondary end points were at the favor of Radium-223 treated patients, including time to first skeletal related event, quality of life and various biochemical end points. However, patient reported pain scores were not collected in the trial. Radium-223 treatment was well tolerated, with the most prominent side effects (all grades) thrombocytopenia 12 and 6%, neutropenia 5 and 1% and diarrhea 25 and 15% in the Radium-223 and placebo arm, respectively.

A post-hoc analysis showed an equal efficacy of Radium-223 treatment in docetaxel pre-treated patients as in docetaxel naïve patients.

In this registry the investigators aim to evaluate the efficacy of Radium-223 treatment and first subsequent therapy in a non-study population. Various parameters will be collected, including changes in patient reported pain score. Moreover, changes in serum and blood levels of biomarkers of bone metabolism and levels of blood osteoclast precursors in Radium-223 treated patients will be evaluated for their potential to predict treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

* At the physicians discretion

Exclusion Criteria:

* At the physicians discretion
* Radium-223 treatment in combination with another life-prolonging agent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastasized castration resistant prostate cancer (mCRPC), who have bone metastases and no visceral metastases and receive Radium-223 according to the physician's discretion
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2015-01-17 (Actual); Primary Completion 2015-02-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Reported analgesic use and pain outcome | through study completion, an average of 1 year. (6 months treatment, 6 months follow-up after end of treatment)
  Evaluate Radium-223 treatment efficacy by patient reported analgesic use and pain outcome, assessed by BPI-S, FACT-P and questionnaire about analgesic use.

SECONDARY OUTCOMES:
Efficacy on clinical parameters of treatment with Radium-223 | through study completion, an average of 1 year. (6 months treatment, 6 months follow-up after end of treatment)
  Evaluate Radium-223 treatment efficacy in a non-study population of CRPC patients by clinical parameters, through patient records (WHO PS)
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | through study completion, an average of 1 year. (6 months treatment, 6 months follow-up after end of treatment)
  Evaluate Radium-223 treatment tolerability in a non-study population of CRPC patients, through patient records (using the CTCAE v4.03 for adverse events).
Subsequent therapy after Radium-223: Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | through study completion, an average of 1 year. (6 months treatment, 6 months follow-up after end of treatment)
  Evaluate of the treatment after Radium-223 the treatment tolerability in a non-study population of CRPC patients, through patient records (using the CTCAE v4.03 for adverse events).
Efficacy of subsequent treatment on clinical parameters | through study completion, an average of 1 year. (6 months treatment, 6 months follow-up after end of treatment)
  Evaluate the subsequent treatment efficacy in a non-study population of CRPC patients by clinical parameters, through patient records (WHO PS) But also by patient records (recors of bonescans, CT scans, blood measurements, out-patient clinic visits).
Symptomatic Skeletal Events | through study completion, an average of 1 year. (6 months treatment, 6 months follow-up after end of treatment)
  To evaluate the efficacy of Radium-223 treatment in a nonstudy population by effects on Symptomatic Skeletal Event (SSE). Through patient records and questionnairs (FACT-P, BPI-S and use of painmedication)
Evaluate the efficacy of Radium-223 by patient records | through study completion, an average of 1 year. (6 months treatment, 6 months follow-up after end of treatment)
  Records of bonescans, CT scans, blood measurements, this will all be combined in one reported value; Progressve disease, stable disease, partial remission or complete remission.

CONTACTS AND LOCATIONS:
Overall Officials: Andre Bergman, MD, PhD, Principal Investigator — The Netherlands Cancer Institute
Locations (20):
- Netherlands (20):
  - Meander Medical Center, Amersfoort, Utrecht
  - Jeroen Bosch Hospital, 's-Hertogenbosch
  - Noordwest Ziekenhuisgroep, Alkmaar
  - Zorggroep Twente, Almelo
  - The Netherlands Cancer Intitute, Amsterdam
  - Rijnstate, Arnhem
  - Amphia Ziekenhuis, Breda
  - Reinier de Graaf Hospital, Delft
  - Deventer Ziekenhuis, Deventer
  - Catharina Ziekenhuis, Eindhoven
  - Groene Hart Ziekenhuis, Gouda
  - Martini Ziekenhuis, Groningen
  - Atrium Medisch Centrum Parkstad, Heerlen
  - Spaarne Gasthuis, Hoofddorp
  - Antonius Ziekenhuis, Nieuwegein
  - Franciscus Gasthuis-Vlietland, Rotterdam
  - Haga Ziekenhuis, The Hague
  - MC Haaglanden, The Hague
  - Universitair Medisch Centrum Utrecht, Utrecht
  - Isala Klinieken, Zwolle